CLINICAL TRIAL: NCT01301482
Title: Ear Acupuncture for Acute Sore Throat in Patients Unable to Take Non-steroidal Anti-inflammatory Agents (NSAIDs)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study is no longer necessary (outmoded, outdated, science has changed)
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FWH20110009H
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Acute Sore Throat
Keywords: Acute Sore Throat; Ear Acupuncture
MeSH Terms: interventions — Acupuncture, Ear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- battlefield auricular acupuncture (Experimental)
  Interventions: Device: Ear Acupuncture
- placebo (No Intervention)

INTERVENTIONS:
Device: Ear Acupuncture — Ear acupuncture utilizes up to 10 needles (see figure 6). If at any point the subject decides not to continue with the placing of the needles, the acupuncture will cease and the number of points will be documented. The ear Acupuncture points on the right ear include Cingulate gyrus, thalamus, omega 2, shen-men, point zero. The ear Acupuncture points on the left ear include Cingulate gyrus, thalamus, omega 2, shen-men, point zero (see figures 1-5).
  Arms: battlefield auricular acupuncture

SUMMARY:
The purpose of this study is to assess the effect of ear acupuncture alone in subjects with a contraindication to anti-inflammatory medications in the reduction of pain and hours lost from work in acute sore throat.

ELIGIBILITY:
Inclusion:

* Male and female subjects (DoD beneficiaries), 18 years or older, with upper respiratory complaints and their primary symptom being acute sore throat.
* Minimum pain score of 5 points on a 11 point scale (0-10 with 10 being the worst pain)

The above with any one of the following:

* Allergy to Non-Steroidal Anti-inflammatory agents (NSAIDs)
* History of significant gastrointestinal bleed
* Previous documented history of stage 2 kidney disease or worse
* History of gastric bypass surgery
* Chronic oral steroids use

Exclusion:

* Absence of one or more ears
* Known Pregnancy
* Known Peritonsillar abscess (PTA)
* Throat, mouth or esophageal cancer
* Active cellulitis of ear
* Ear anatomy precluding identification of acupuncture landmarks
* Use of Hearing Aids that preclude the use of ear acupuncture
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Moss, M.D., Principal Investigator — Mike O'Callaghan Federal Hospital/Nellis Air Force Base
Locations (1):
- Mike O'Callaghan Federal Hosptial, Nellis Air Force Base, Nevada, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was terminated after 3 subjects were recruited. Study was no longer necessary (outmoded, outdated, science has changed)
Period: Overall Study
Arm/Group | Battlefield Auricular Acupuncture
Started | 3
Completed | 2
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Battlefield Auricular Acupuncture: This single arm study places ear acupuncture needles alone in patients reporting acute sore throat and to whom NSAIDs are a contraindication.
  Ear Acupuncture: Ear acupuncture utilizes up to 10 needles. If at any point the subject decides not to continue with the placing of the needles, the acupuncture will cease and the number of points will be documented. The ear Acupuncture points on the right ear include Cingulate gyrus, thalamus, omega 2, shen-men, point zero. The ear Acupuncture points on the left ear include Cingulate gyrus, thalamus, omega 2, shen-men, point zero.
Arm/Group | Battlefield Auricular Acupuncture
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
sore throat culture taken [Count of Participants; unit: Participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Pain on Numeric Pain Rating Scale
Description: Does ear acupuncture alone significantly reduce pain in acute sore throat? Measured by reduction in pain on 0-10 (10 highest pain) numeric pain rating scale.
Time Frame: initial, 15 minute post, 6 hours post, 24 hours post, 48 hours post
Population: Study was terminated. Any data collected could not be meaningfully reported. Here we report initial data collected before study termination.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Battlefield Auricular Acupuncture
Number analyzed (Participants) | 3
units on a scale
  initial pain | 6 [5 to 7]
  pain 15 minutes post battlefield acupuncture | 1.7 [0 to 4]
  pain 6 hours post battlefield acupuncture | 1.7 [1 to 2]
  pain 24 hours post battlefield acupuncture | 1 [0 to 2]
  pain 48 hours post battlefield acupuncture: number analyzed (Participants) | 2
  pain 48 hours post battlefield acupuncture | 0 [0 to 0]

ADVERSE EVENTS:
Groups:
- Battlefield Auricular Acupuncture: There were 0 adverse events of any severity. Study was terminated as no longer necessary (outmoded, outdated, science has changed)
Arm/Group | Battlefield Auricular Acupuncture
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
Study was terminated after three subjects were recruited. 33 were predicted in protocol to be enough to analyze meaningful data, alas, only 3 were recruited. Study was no longer necessary (outmoded, outdated, science has changed)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes